CLINICAL TRIAL: NCT06327152
Title: Caffeine Use in the Management of Preterm Infants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Cherry Uy, HS Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2659
Record Dates: First submitted 2024-03-13; First posted 2024-03-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Apnea of Prematurity
Keywords: Feeding; Caffeine
MeSH Terms: conditions — Apnea | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blinded, placebo-controlled trial of 40 preterm infants born at less than or equal to 32 weeks and 0 days gestation. Infants will be randomized to receive either caffeine or placebo for up to maximum of additional four (4) weeks after meeting clinical criteria to come off caffeine.
Who Masked: Participant, Investigator
Masking Description: Families, nurses, therapists, and doctors will be blinded. Only pharmacy will be unblinded and know which subjects are in each treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caffeine Group (Active Comparator): Infants randomized to receive caffeine will continue to receive caffeine at standard of care maintenance dose of 10-15 mg/kg/day given every 24 hours. The dose will be weight adjusted every 7 days, starting on the day of enrollment. Caffeine will be given enterally, via nasogastric tube or by mouth.
  Interventions: Drug: Caffeine
- Placebo Group (Placebo Comparator): Infants randomized to the placebo group will be given sterile water at an equivalent volume to the volume if caffeine were to be given, using the previous weight-based caffeine dose. The placebo will be given every 24 hours. The dose/volume will be weight adjusted every 7 days, starting on the day of enrollment. The placebo will be given enterally, via nasogastric tube or by mouth.
  Interventions: Other: Sterile Water Placebo

INTERVENTIONS:
Drug: Caffeine — Infants randomized to receive caffeine will continue to receive caffeine at the current weight-based dose (which is the standard of care maintenance dose of 10-15 mg/kg/day) given every 24 hours. The weight-based dose calculated using the weight at the time of enrollment will be the weight-based dose used for the duration of the study. The dose will be weight adjusted every 7 days, starting on the day of enrollment. Caffeine will be given enterally, via nasogastric tube or by mouth.
  The study drug (caffeine) will be administered for a maximum of 4 weeks. The study drug will be discontinued after 4 weeks or when the infant reaches Step 4 of our institution's oral feeding protocol (oral feeding 6 times per day), whichever comes first. The study drug will also be discontinued if the open-label maintenance caffeine is started by the clinical team based on clinical indications.
  Arms: Caffeine Group
Other: Sterile Water Placebo — Infants randomized to the placebo group will be given sterile water at an equivalent volume to the volume if caffeine were to be given, using the previous weight-based caffeine dose. The placebo will be given every 24 hours. The dose/volume will be weight adjusted every 7 days, starting on the day of enrollment. The placebo will be given enterally, via nasogastric tube or by mouth.
  The placebo will be administered for a maximum of 4 weeks. The placebo will be discontinued after 4 weeks or when the infant reaches Step 4 of our institution's oral feeding protocol (oral feeding 6 times per day), whichever comes first. The placebo will also be discontinued if the open-label maintenance caffeine is started by the clinical team based on clinical indications.
  Arms: Placebo Group

SUMMARY:
This study aims to assess whether extending the duration of caffeine therapy will help preterm infants achieve full oral feeding faster.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo-controlled trial. Infants will be randomized to receive either caffeine or placebo for up to maximum of four additional weeks after meeting clinical criteria to discontinue caffeine. Initiation of oral feeding will be based on standard of care as determined by a neonatal occupational therapist and clinical cues. Oral feedings will be advanced by a standardized 5 step oral feeding protocol. The time it takes to achieve full oral feeds between the treatment and control groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

• Infants born at equal to or less than 32 weeks and 0 days gestational age AND

* Equal to or greater than 34 weeks and 0 days corrected gestation at time of enrollment.
* Off respiratory support for at least 2 days (nasal canula oxygen, high flow nasal canula, continuous positive airway pressure (CPAP), mechanical ventilation).
* On caffeine and meet criteria to discontinue caffeine.
* No significant cardiopulmonary events for at least 5 days (apnea > 20 seconds, apnea with heart rate (HR) < 80 beats per minute (bpm), HR < 80 bpm with desaturation < 85% or color change).

Exclusion Criteria:

* Infants with critical congenital heart disease.
* Infants with neuromuscular conditions affecting respiration.
* Infants with overt brain injury (i.e. severe Grade 3-4 intraventricular hemorrhage, cystic periventricular leukomalacia) that may affect oral feeding.
* Infants with major genetic disorders.
* Infants with anatomic anomalies that will hinder oral feeding.
* Infants who have already progressed to Step 3 (of 5) of our institution's oral feeding protocol (oral feeds 4 times per day).
* Infants who develop necrotizing enterocolitis after enrollment.
* Failure to obtain consent or declined by parents.

Ages: 1 Week to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to full feeds | From first nutritive oral feed until full oral feeds achieved, up to 6 weeks
  The primary outcome is time (in days) to full oral bottle feeding or breastfeeding or a combination of both. Full oral bottle feeding is defined as 48 hours of consistent intake of at least 150ml/kg/day of formula or breastmilk. If the subject is on combination of bottle and breastfeeding, two consecutive days of positive weight gain will be used in place of 150ml/kg/day as primary outcome measure.

SECONDARY OUTCOMES:
Time to discharge | Randomization until discharge, up to 6 weeks
  Time to discharge measured in days of hospitalization after randomization
Post menstrual age (PMA) at time of discharge | Randomization until discharge, up to 6 weeks
  Post menstrual age at discharge
Number of significant cardiopulmonary events | Randomization until discharge, up to 6 weeks
  Number of significant cardiopulmonary events defined as apnea > 20 seconds, apnea with heart rate (HR) < 80 beats per minute (bpm), HR < 80 bpm with desaturation < 85% or color change. Significant events are ones that occur while infant is asleep or lying down.
Weight change | Randomization until discharge, up to 6 weeks
  Weight change measured by change in grams

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Uy, MD, Principal Investigator — UC Irvine
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No